CLINICAL TRIAL: NCT03719781
Title: Postoperative Cognitive Dysfunction in Patients Undergoing Pituitary Removal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Cennet Tor Kılıc, Anesthesiology and Reanimation Resident, Kocaeli University
Other Study IDs: GOKAEK 2017/153
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Pituitary Tumor
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group1: patients undergoing pituitary tumor removal surgery will be tested with standardized minimental testing.
  Interventions: Diagnostic Test: standardized minimental testing

INTERVENTIONS:
Diagnostic Test: standardized minimental testing — To diagnose postoperative cognitive dysfunction

SUMMARY:
As postoperative cognitive dysfunction rates are high especially in elder patients, cognitive dysfunction is not diagnosed and treated effectively. This statement is associated with prolonged hospital stays by increasing morbidity. We wanted to see the incidency of postoperative cognitive dysfunction in patients undergoing elective pituitary tumor removal surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Undergoing elective pituitery tumor removal surgery

Exclusion Criteria:

* >II ASA scores
* Using antidepressant agents
* Patient refusal
* Mental diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Undergoing elective pituitary tumor removal surgery
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
minimental test score | preoperative 24th hour
  scores between 0-30
minimental test score | postoperative 4th hour
  scores between 0-30
minimental test score | postoperative 24th hour
  scores between 0-30
minimental test score | one month after discharged
  scores between 0-30

CONTACTS AND LOCATIONS:
Overall Officials: Cennet Tor Kılıç, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No